CLINICAL TRIAL: NCT01896544
Title: The Effect of Cholecalciferol Supplementation on Vitamin D Status in Sepsis
Brief Title: Cholecalciferol Supplementation for Sepsis in the ICU
Acronym: CSI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Sadeq A. Quraishi, Assistant Professor of Anaesthesia, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2013P001406
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Results first posted 2016-06-13 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-05

CONDITIONS: Hypovitaminosis D
Keywords: cholecalciferol; vitamin D; sepsis; infection
MeSH Terms: conditions — Vitamin D Deficiency; Sepsis; Infections | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cholecalciferol Dose II (Active Comparator): Oral suspension cholecalciferol 400,000 IU
  Interventions: Dietary Supplement: Cholecalciferol
- Placebo (Placebo Comparator): Oral suspension of placebo cholecalciferol
  Interventions: Dietary Supplement: Placebo
- Cholecalciferol Dose I (Active Comparator): Oral suspension cholecalciferol 200,000 IU
  Interventions: Dietary Supplement: Cholecalciferol

INTERVENTIONS:
Dietary Supplement: Cholecalciferol — 7ml syringe of cholecalciferol suspension given through nasogastric (NG) or orogastric (OG) tube
  Arms: Cholecalciferol Dose I; Cholecalciferol Dose II
Dietary Supplement: Placebo — 7ml syringe of placebo cholecalciferol suspension given through nasogastric (NG) or orogastric (OG) tube
  Arms: Placebo

SUMMARY:
Sepsis in a clinical entity that occurs in patients with serious infections. Though the severity of illness may vary, every year, approximately 1.6 million Americans are treated for sepsis. Even with timely interventions, anywhere from 16% to >80% of patients with sepsis will not survive. Immune dysfunction is thought to play a critical role in the ability for infections to evolve into sepsis and to eventually lead to death. Recently, vitamin D has been identified as a key regulator of the immune system. While it remains unclear whether optimizing vitamin D status may improve outcomes in sepsis, little is known about the effects of vitamin D supplementation in patients with severe infections. As such, our goal is to study whether high doses of cholecalciferol (vitamin D3) can improve vitamin D status and boost certain aspects of the immune system in patients with sepsis.

DETAILED DESCRIPTION:
Sepsis is a clinical syndrome that complicates severe infections. It is characterized by the cardinal signs of inflammation (e.g. vasodilation, leukocytosis, increased microvascular permeability) occurring in tissues that are remote from the site of an infection. Current theories about the onset and progression of the sepsis syndrome focus on dysregulation of inflammatory responses, including the possibility that a massive and uncontrolled release of pro-inflammatory mediators initiates a chain of events that lead to widespread tissue injury. The degree of immune dysfunction is thought to correlate with the severity of the sepsis syndrome. Sepsis syndrome can range from sepsis, to severe sepsis, septic shock, and multiple organ dysfunction syndrome (MODS). The mortality associated with each of these is estimated to be 16%, 20%, 46%, >80%, respectively. The annual incidence of sepsis syndrome exceeds 1.6 million cases in the United States alone.

Recently, cells of the innate and adaptive immune system have been shown to express the vitamin D receptor. Vitamin D appears to be necessary for interferon-γ dependent T cell responses to infection. In low vitamin D states, dysfunctional macrophage activity becomes evident. Vitamin D is also an important link between Toll Like Receptor (TLR) activation and antibacterial response. Human macrophages stimulated by TLR induce: 1) vitamin D receptor expression; 2) conversion of 25(OH)D to its most biologically active form of 1,25-dihydroxyvitamin D; and 3) production of cathelicidin (LL-37), an endogenous antimicrobial peptide with potent activity against bacteria, viruses, fungi, and mycobacteria. LL-37 is highly expressed in both the plasma and at natural barrier sites (e.g. skin, gut, lungs) and may represent an important first-line of defense for the innate immune system.

In humans, cholecalciferol (vitamin D3) is either obtained through the diet or synthesized by skin upon exposure to ultraviolet B (UVB) radiation. Cholecalciferol is converted to 25(OH)D in the liver or by cells of the immune system. Serum 25(OH)D can be measured with relative ease and is the most abundant vitamin D metabolite. It is therefore, often used as a proxy for total body vitamin D status and 25(OH)D levels <30 ng/mL characterize an insufficient state. A growing body of evidence suggests that a significant proportion (50-90%) of critically ill patients may have insufficient 25(OH)D levels during admission to the intensive care unit (ICU). 25(OH)D insufficiency, in turn, appears to be associated with a higher risk of mortality in critically ill patients. However, randomized, placebo-controlled trials (RCTs) aimed at studying the effect of vitamin D supplementation in critical illness are limited and have largely focused on superficial assessments of vitamin D status. While it is known that septic patients have nearly universally low 25(OH)D levels and that the vitamin D levels are inversely correlated with the severity of sepsis, little is known regarding the effects of vitamin supplementation in this patient cohort. Therefore, our goal is to determine whether vitamin D supplementation in patients highly suspected of sepsis syndrome may be effective in optimizing 25(OH)D levels and in improving host production of the antimicrobial polypeptide LL-37.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking
* Within 24 hours of a suspected diagnosis of sepsis
* Meeting criteria for sepsis (defined as suspected or confirmed infection AND at least one diagnostic criteria in each of the following groupings):

  1. Vital signs:

     1. Temperature: >38.3 Celsius (C) or <36 Celsius (C)
     2. Heart rat e: >90/min, or >2 standard deviation above normal
     3. Tachypnea (>20 breaths per minute)
     4. Altered mental status
     5. Positive fluid balance (>20 mL/Kg over 24 hrs)
     6. Glucose >140 mg/dL in the absence of diabetes mellitus
  2. Inflammatory markers:

     1. white blood cell (WBC): >12,000 or <4,000
     2. Normal WBC count with >10% immature forms
     3. c-reactive protein (CRP) >2 standard deviation above normal value
     4. Pro- calcitonin >2 standard deviation above normal value
  3. Hemodynamic

     1. Systolic blood pressure (SBP) <90 millimeters mercury (mmHg), Mean Arterial Pressure (MAP) <70mmHg or SBP decrease >40mmHg
     2. Vasopressor therapy to maintain MAP >65mmHg
  4. Organ dysfunction

     1. Arterial hypoxemia arterial oxygen partial pressure/fractional inspired oxygen (PaO2/FiO2) <300
     2. Acute Oliguria (UoP <0.5 mL/Kg/hr for at least 2 hours)
     3. Cr increase >0.5 mg/dL
     4. Coagulopathy: internationals normalized ratio (INR) >1.5 or a-partial prothrombin time (aPTT) >60 sec
     5. Thrombocytopenia: Platelet (PLT) <100 thousand (K)
     6. Hyperbilirubinemia: Total Bilirubin (Tbili) >4 mg/dL
  5. Tissue perfusion

     1. Lactate >2 mmol/L
     2. Decrease cap refill or mottling

Exclusion Criteria:

* Pregnant females or immediate post-partum status
* "Comfort measures only" status
* Inability to provide informed consent or have a surrogate consent
* History of renal stones within the past year
* History of hypercalcemia within the past year
* Baseline serum total calcium >10 mg/dL
* Established diagnosis associated with increased risk of hypercalcemia (e.g. metastatic cancer, sarcoidosis, multiple myeloma, primary hyperparathyroidism)
* History of severe anemia (Hematocrit <25%)
* Medications that affect vitamin D metabolism (e.g. antiepileptics, tuberculosis medication
* Already enrolled or planning to enroll in a research study that would conflict with full participation in the current study or confound the observation or interpretation of the study findings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sadeq A Quraishi, MD, MHA, MMSc, Principal Investigator — Harvard Medical School, Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Oral suspension of placebo cholecalciferol
  Placebo: 7ml syringe of placebo cholecalciferol suspension given through NG or OG tube
- Cholecalciferol Dose I: Oral suspension cholecalciferol 200,000 IU
  Cholecalciferol: 7ml syringe of cholecalciferol suspension given through NG or OG tube
- Cholecalciferol Dose II: Oral suspension cholecalciferol 400,000 IU
  Cholecalciferol: 7ml syringe of cholecalciferol suspension given through NG or OG tube
Period: Overall Study
Arm/Group | Placebo | Cholecalciferol Dose I | Cholecalciferol Dose II
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cholecalciferol Dose II | Placebo | Cholecalciferol Dose I | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [59 to 67] | 65 [58 to 70] | 64 [55 to 66] | 64 [58 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 4 | 12
  Male | 6 | 6 | 6 | 18
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 30
Body mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 30 [28 to 37] | 28 [26 to 35] | 28 [27 to 33] | 28 [27 to 33]
Acute Physiology and Chronic Health Evaluation II (APACHE II) score [Median (Inter-Quartile Range); unit: scores on a scale] — The APACHE II score is a severity-of-disease classification used in the intensive care unit. The APACHEII score is calculated within within 24 hours of admission. Higher scores correspond with more severe disease and therefore increased risk of death. The score ranges from 0-71 points.
  scores on a scale | 23 [16 to 25] | 22 [16 to 28] | 21 [19 to 32] | 22 [16 to 28]
Intensive Care Unit (ICU) type [Number; unit: participants]
  medical | 5 | 6 | 5 | 16
  surgical | 5 | 4 | 5 | 14
Positive culture [Number; unit: percentage] — Totals do not equal 100% since some patients had more than one location where a positive culture was obtained.
  percentage
    Pulmonary | 40 | 40 | 50 | 130
    Blood stream | 70 | 60 | 60 | 190
    Urinary | 10 | 10 | 10 | 30
Day 1 data: 25 hydroxyvitaminD(25OHD),bioavailable 25 hydroxyvitamin D(B25OHD), cathelicidin (LL-37) [Median (Inter-Quartile Range); unit: ng/mL]
  Day 1 25OHD (ng/mL) | 17 [13 to 25] | 19 [13 to 22] | 15 [12 to 20] | 17 [13 to 22]
  Day 1 B25OHD (ng/mL) | 2.5 [1.7 to 2.9] | 1.4 [0.8 to 2.1] | 1.9 [1.2 to 2.5] | 1.9 [1.2 to 2.1]
  Day 1 LL-37 (ng/mL) | 51 [41 to 52] | 53 [43 to 62] | 52 [48 to 59] | 52 [43 to 59]
30 day readmission [Number; unit: participants]
  No | 10 | 8 | 10 | 28
  Yes | 0 | 2 | 0 | 2
30 day mortality [Number; unit: participants]
  dead | 2 | 3 | 3 | 8
  alive | 8 | 7 | 7 | 22
Day 1 data: high-sensitivity c-reactive protein (hs-CRP) [Median (Inter-Quartile Range); unit: mg/L] | 119 [85 to 247] | 106 [60 to 267] | 208 [90 to 359] | 119 [85 to 267]
Day 1: total body fluid balance (TBB) [Median (Inter-Quartile Range); unit: mL] | 1,518 [696 to 2,088] | 1592 [1,086 to 2,117] | 1,730 [925 to 3075] | 1,592 [925 to 2,117]

OUTCOME MEASURES:

1. Primary Outcome: Change in Vitamin D Status 5 Days Following Supplementation With Cholecalciferol
Description: Subjects will receive 200,000 IU or 400,000 IU cholecalciferol suspension (vs. placebo) within 24 hours from the onset of a suspected case of sepsis during their hospitalization. Vitamin D status at the onset of a suspected case of sepsis will be compared to vitamin D status between 5-9 days after supplementation with cholecalciferol or placebo. To assess vitamin D status, we will measure serum and urine: 1) 25-hydroxyvitamin D; 2) 1,25-dihydroxyvitamin D; 3) 24,25-dihydroxyvitamin D; 4) Fibroblast growth factor 23; 5) Vitamin D binding protein; 6) LL-37; 7) Parathyroid hormone; 8) Albumin; 9) Calcium; and 10) Phosphorus levels.
Time Frame: Patients will be followed between the onset of suspected sepsis and for an average duration of 7 days
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Placebo | Cholecalciferol Dose I | Cholecalciferol Dose II
Number analyzed (Participants) | 10 | 10 | 10
ng/mL
  Day 1 | 19 [13 to 22] | 15 [12 to 20] | 17 [13 to 25]
  Day 5 | 19 [11 to 23] | 22 [16 to 25] | 29 [23 to 41]

2. Secondary Outcome: Change in Immunological Profile 5 Days Following Supplementation With Cholecalciferol
Description: Subjects will receive 200,000 IU or 400,000 IU cholecalciferol suspension (vs. placebo) within 24 hours from the onset of a suspected case of sepsis during their hospitalization. Immunological profile at the onset of a suspected case of sepsis will be compared to the immunological profile between 5-9 days after supplementation with cholecalciferol or placebo. To assess the immunological profile, we will measure serum LL-37.
Time Frame: Patients will be followed between the onset of suspected sepsis and for an average duration of 7 days
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Placebo | Cholecalciferol Dose I | Cholecalciferol Dose II
Number analyzed (Participants) | 10 | 10 | 10
ng/mL
  Day 1 LL-37 (ng/mL) | 53 [43 to 62] | 52 [48 to 59] | 51 [41 to 52]
  Day 5 LL 37 (ng/mL) | 50 [35 to 54] | 54 [40 to 64] | 67 [59 to 68]

3. Secondary Outcome: Incidence of Infection-related Complications Within 90 Days From the Onset of a Suspected Case of Sepsis
Description: Subjects will receive 200,000 IU or 400,000 IU cholecalciferol suspension (vs. placebo) within 24 hours from the onset of a suspected case of sepsis during their hospitalization. The incidence of infection-related complications will be assessed between the onset of suspected sepsis and 80-100 days after supplementation with cholecalciferol or placebo. To assess the incidence of infection-related complications, we will measure rates of: 1) ICU length of stay; and 2) hospital length of stay
Time Frame: Patients will be followed between the onset of suspected sepsis and for an average duration of 90 days
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Cholecalciferol Dose I | Cholecalciferol Dose II
Number analyzed (Participants) | 10 | 10 | 10
days
  ICU length of stay | 12 [7 to 15] | 4 [3 to 11] | 3 [2 to 11]
  Hospital length of stay | 21 [18 to 31] | 13 [12 to 16] | 14 [8 to 21]

4. Secondary Outcome: Incidence of Infection-related Complications Within 90 Days From the Onset of a Suspected Case of Sepsis
Description: Subjects will receive 200,000 IU or 400,000 IU cholecalciferol suspension (vs. placebo) within 24 hours from the onset of a suspected case of sepsis during their hospitalization. The incidence of infection-related complications will be assessed between the onset of suspected sepsis and 80-100 days after supplementation with cholecalciferol or placebo. To assess the incidence of infection-related complications, we will measure rates of:
  1) 30 day hospital readmission; and 2) 30 day mortality.
Time Frame: Patients will be followed between the onset of suspected sepsis and for an average duration of 90 days
Measure: Number; unit: participants
Arm/Group | Placebo | Cholecalciferol Dose I | Cholecalciferol Dose II
Number analyzed (Participants) | 10 | 10 | 10
participants
  30 day readmission: no | 8 | 10 | 10
  30 day readmission: yes | 2 | 0 | 0
  30 day mortality: dead | 3 | 3 | 2
  30 day mortality:alive | 7 | 7 | 8

5. Secondary Outcome: Change in Immunological Profile 5 Days Following Supplementation With Cholecalciferol
Description: Subjects will receive 200,000 IU or 400,000 IU cholecalciferol suspension (vs. placebo) within 24 hours from the onset of a suspected case of sepsis during their hospitalization. Immunological profile at the onset of a suspected case of sepsis will be compared to the immunological profile between 5-9 days after supplementation with cholecalciferol or placebo. To assess the immunological profile, we will measure serum hsCRP.
Time Frame: Patients will be followed between the onset of suspected sepsis and for an average duration of 90 days
Measure: Median (Inter-Quartile Range); unit: mg/L
Groups:
- Cholecalciferol Dose 1: Oral suspension cholecalciferol 200,000 IU
- Cholecalciferol Dose 2: Oral suspension of cholecalciferol 400,000 IU
Arm/Group | Placebo | Cholecalciferol Dose 1 | Cholecalciferol Dose 2
Number analyzed (Participants) | 10 | 10 | 10
mg/L
  Day 1 hsCRP (mg/L) | 106 [60 to 267] | 208 [90 to 369] | 119 [85 to 247]
  D 5 hsCRP (mg/L) | 53 [38 to 72] | 98 [12 to 130] | 31 [26 to 160]

ADVERSE EVENTS:
Time Frame: Time frame for Adverse Event was until study completion, until the 7th day of study participation
Description: Serious and Other Adverse Events were monitored for the placebo arm but none were observed.
Arm/Group | Placebo | Cholecalciferol Dose I | Cholecalciferol Dose II
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No